CLINICAL TRIAL: NCT06596278
Title: Development of Memesto, a Wearable Repetitive Message and Music Therapy Device That Senses and Reduces Agitation in Persons With AD/ADRD
Brief Title: Memesto Wearable Repetitive Message and Music Therapy Device Music Therapy Device That Senses and Reduces Agitation in People With AD,
Acronym: AWARD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Edgewater Safety Systems, Inc. (Industry)
Collaborators: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Jeffery T. Banker, President, Edgewater Safety Systems, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: ESS-MEM-001
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Alzheimer's Disease
Keywords: dementia; Alzheimer's disease
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Intervention Model Description: Stage 1
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Memesto Intervention (Experimental): Memesto device intervention
  Interventions: Device: Memesto

INTERVENTIONS:
Device: Memesto — Memesto wearable audio player

SUMMARY:
This is a 12-week proof-of-concept study to evaluate the efficacy of Memesto in reducing agitation in persons with Alzheimer's disease and Alzheimer's disease related dementias (AD/ADRD) currently living in a residential care facility. It is hypothesized that Memesto use will result in a reduction in agitation.

DETAILED DESCRIPTION:
After informed consent is obtained and preliminary eligibility established, participants will be trained and issued the Memesto device for use over a 2-week screening/training phase. Participants successfully completing this phase will proceed into a 10-week open label treatment phase (via telephone and/or in-person data collection).

ELIGIBILITY:
Inclusion Criteria: Given that people living with ADRD can be of any adult age, people meeting criteria for ADRD diagnosis will be regardless of age. Younger-onset people living with ADRD, which may be smaller, will be considered for participation along with adults older than age 65 that make up the largest portion of persons living with ADRD. The family and professional caregivers can be any age greater than eighteen. We anticipate that 5% of the People living with ADRD will be less than age 65 with 70% being greater than age 75 and 25% being between ages 65 and 74. For family caregivers, we envision most will be spouses with the same age distributions as the parents with a skew to a slightly younger age group for caregivers who are children of the person living with ADRD and/or the spouses of children. For professional caregivers, we anticipate they will be between the residential care workforce ages of 20 and 65 with a skew toward persons over age 40.

Inclusion/Exclusion Criteria: Eligible participants will be adults with a dementia diagnosis who have clinically significant agitation, defined as a state of poorly organized and purposeless psychomotor activity characterized by at least one of the following: aggressive verbal (screaming, cursing), aggressive physical (destroying objects, grabbing, fighting), or non-aggressive physical (restlessness, pacing) behaviors. The behavioral symptoms must be severe enough to warrant pharmacological treatment. A family caregiver must be willing to participate along with a professional caregiver from the resident living facility.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-11-21 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Average score on the Neuropsychiatric Inventory (NPI) agitation domain | 10 weeks
  The scores on the NPI agitation domain at baseline will be the comparator. A score of zero indicates no agitation is observed. If agitation is mentioned, caregivers will rate the agitation symptom frequency from 1 to 4 (less than once a week, about one time a week, several times a week, or more than once per day). Severity for each symptom is rated from 1 to 3 (mild, moderate, or marked). The NPI's composite (frequency x severity) score ranges from 1 to 12 for each positively endorsed domain.13 The average of the family and professional caregiver rating will be utilized

CONTACTS AND LOCATIONS:
Overall Officials: Raj C. Shah, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush Alzheimer's Disease Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
The data will be made available on the Rush Alzheimer's Disease Center Research Resource Sharing Hub, which has descriptions of the studies and variables. It has a dynamic query function to aid searches for data. Researchers can set up a login account and then submit requests for data by following the instructions. Data Use Agreements are available for download. A request for data will be sent to Dr. Raj Shah (site PI for the study) via automated email alert that a request has been submitted. This initiates a web-based review process with regular and ad hoc reviewers to include a representative from Edgewater chosen based on required expertise. Upon approval and signature of a data use agreement, the data will be shared with the requestor. All requests, reviews, electronic discussions, and the final disposition of each request are archived.
Supporting Information: Study Protocol, ICF
Time Frame: Sharing of data is planned at the time of publication of the primary results or within 9 months of database lock, whichever comes first.
Access Criteria: Researchers can set up a login account and then submit requests for data by following the instructions. Data Use Agreements are available for download. A request for data will be sent to Dr. Raj Shah (site PI for the study) via automated email alert that a request has been submitted. This initiates a web-based review process with regular and ad hoc reviewers to include a representative from Edgewater chosen based on required expertise. Upon approval and signature of a data use agreement, the data will be shared with the requestor. All requests, reviews, electronic discussions, and the final disposition of each request are archived.

DOCUMENTS (2):
  • Study Protocol (2021-12-01): https://cdn.clinicaltrials.gov/large-docs/78/NCT06596278/Prot_000.pdf
  • Informed Consent Form (2021-12-30): https://cdn.clinicaltrials.gov/large-docs/78/NCT06596278/ICF_001.pdf